CLINICAL TRIAL: NCT01141777
Title: The Effects of Spirulina Platensis on Insulin Resistance in HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Collaborators: University of Yaounde (Other); Antenna Technologies (Unknown)
Responsible Party: Dr Sobngwi Eugene, Consultant Endocrinologist and Senior Lecturer, University of Yaounde 1, Cameroon and Newcastle University, UK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MAK-GLE_Spirulina
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-09

CONDITIONS: Insulin Resistance; HIV/AIDS
Keywords: Spirulina platensis; Insulin resistance; HIV/AIDS; HAART; Soya beans
MeSH Terms: conditions — Insulin Resistance; Acquired Immunodeficiency Syndrome | interventions — Soybean Oil; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spirulina platensis (Active Comparator)
  Interventions: Dietary Supplement: Spirulina platensis
- Soya bean (Placebo Comparator)
  Interventions: Dietary Supplement: Soya bean

INTERVENTIONS:
Dietary Supplement: Spirulina platensis — Subjects received 19g daily of supplement averagely.This was supplied as powder daily, in packs that lasted for 2weeks each. Each subject was therefore seen every two week to obtain new stock of supplements and evaluate compliance
  Other Names: Treatment group
  Arms: Spirulina platensis
Dietary Supplement: Soya bean — Each subject received 19g of supplement on average daily. Subjects were seen every two weeks to evaluate compliance and obtain a new stock.
  Other Names: Control group
  Arms: Soya bean

SUMMARY:
Spirulina, a widely used food supplement, improves the lipid profile and glycemic control in people living with diabetes, suggesting that it could have some effects on insulin sensitivity. Since HIV-infected patients develop metabolic abnormalities due to the virus and/or to antiretroviral (ARV) drugs, the investigators therefore proposed to evaluate the effect that spirulina can have on HIV/HAART-associated insulin resistance

DETAILED DESCRIPTION:
Even though antiretroviral therapy (ART) has dramatically improved the health of people living with HIV/AIDS, the prospect of maintaining patients long term on ART can be severely restricted by the development of serious long term effects in their metabolism. These abnormalities include dyslipidemia, lipodystrophy and disorders of glucose metabolism with insulin resistance believed to be the underlying pathophysiological mechanism.

Spirulina, has recently drawn attention on its cholesterol and blood pressure lowering effects, including improvement of glycaemic control in diabetics subjects, suggesting it can have some effects on insulin sensitivity.

The aim of this three month, experimental, prospective, randomised trial was to evaluate the effect of Spirulina on HIV/HAART-associated insulin resistance on 33 subjects. Primary outcome was change in insulin sensitivity during the trial, over two time periods; t=0 and t=12 weeks. The second objective was to compare between the two groups, the percentage of subjects who improved insulin sensitivity by the end of the study.

Recruitment started in October 2008 and the trial ended in February 2009.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection
* Accepted to participate in the study

Exclusion Criteria:

* Acute intercurrent infection
* Treatment that modifies glucose or lipid profile
* Pregnancy
* Known diabetic patient
* Chronic renal failure with calculated creatinine clearance < 60ml/min

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Percentage difference in change in insulin sensitivity between the two groups at the end of eight weeks of intervention | t=0 (baseline), t= week 12 (end of trial)

SECONDARY OUTCOMES:
Percentage of subjects who improved insulin sensitivity by the end of the study, compared between the two groups | t=0 (baseline), t= week 12 (end of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Pr Jean Claude Mbanya, MD, PhD, Study Director — International diabetes federation/ Director, National Obesity Centre, Yaounde Central Hospital, Cameroon; Dr Sobngwi Eugene, MD, PhD, Principal Investigator — Consultant Endocrinologist, National Obesity Centre/ Senior Lecturer, University of Yaounde 1, Cameroon and Newcastle University, UK; Dr Marcel Azabji Kenfack, MD, Study Chair — Dep. of Physiologie, Faculty of Medicine and Biomedical Sciences University Yaoundé I, Cameroon; Dr Gabriel Loni Ekali, MD, Principal Investigator — National Obesity Centre, Yaounde Central Hospital, Cameroon
Locations (1):
- National Obesity Centre, Yaounde Central Hospital, Yaoundé, Centre Region, Cameroon

REFERENCES:
- [Derived] Marcel AK, Ekali LG, Eugene S, Arnold OE, Sandrine ED, von der Weid D, Gbaguidi E, Ngogang J, Mbanya JC. The effect of Spirulina platensis versus soybean on insulin resistance in HIV-infected patients: a randomized pilot study. Nutrients. 2011 Jul;3(7):712-24. doi: 10.3390/nu3070712. Epub 2011 Jul 18. PMID 22254118
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus/
- See also: U.S FDA Resources — http://clinicaltrials.gov/ct2/info/fdalinks